CLINICAL TRIAL: NCT06765785
Title: Cardiovascular Screening in Asymptomatic South Asians - a Pilot Randomized Comparison of Q-risk 3 Score Versus Computed Tomography Coronary Angiography (CTCA)
Brief Title: Cardiovascular Screening in Asymptomatic South Asians
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Vinoda Sharma, Consultant Cardiologist, Sandwell & West Birmingham Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRAS Project ID: 331211
Record Dates: First submitted 2024-12-19; First posted 2025-01-09 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Asymptomatic Condition; South Asian
Keywords: South Asian
MeSH Terms: conditions — Cardiovascular Diseases; Asymptomatic Diseases

STUDY DESIGN:
Intervention Model Description: Pilot randomised study with patients being allocated 1:1 to either Q-risk 3 score or screening CTCA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Q risk 3 score (No Intervention): Q risk 3 score will be calculated and if the 10 year risk of cardiovascular events is >/=10%, patients in this arm will receive primary prevention treatment
- screening CTCA (Experimental): Patients randomised to the CTCA arm will receive primary prevention treatment if plaque is present on the CTCA
  Interventions: Diagnostic Test: CTCA

INTERVENTIONS:
Diagnostic Test: CTCA — Screening CTCA will be performed in the experimental arm after 1:1 randomisation using sealed envelope technique
  Arms: screening CTCA

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of morbidity, mortality and healthcare costs in the United Kingdom. Ethnic minorities like South Asians (SA) have a 3-5 times higher incidence of CVD as predicted by various risk scores despite similar or fewer traditional cardiovascular risk factors.

Computed Tomography Coronary Angiography (CTCA) is able to outline the coronary anatomy determining the site, severity and type of atherosclerotic plaque location in the heart arteries. The National Institute for Health and Care Excellence (NICE) guidelines recommends CTCA as the first line investigation for stable chest pain considered to be coming from the heart (angina).

However there is no pathway for the patients who are asymptomatic but at high risk of CVD, such as the SA cohort. Current practice involves using risk scores to guide management of asymptomatic adults. One recommended and commonly used score is the Q-risk score (the QRISK ® 3-2018 risk calculatorhttps://qrisk.org > three). This score incorporates ethnicity amongst other risk factors and patients with a risk ≥10% of having a heart attack or stroke in the next 10 years are offered primary prevention treatment with low dose statin therapy. For example, an average (height 164cm weight 70kg) 40 year old male of SA descent, without symptoms who is a non-smoker but with Diabetes Mellitus (DM) on tablet treatment scores 5.8% - this risk is not high enough to warrant treatment with a statin unless he also has abnormally raised cholesterol levels. But this patient is still high risk of CVD due to his ethnicity and DM. There is no current evidence to tailor treatment in such asymptomatic, high risk ethnic minorities.

Similar to screening programs for cancer, screening CTCA, compared to risk stratification with the QRISK ® 3 score, may help in risk stratification of a higher proportion of SA patients. 50 asymptomatic SA patients from 2 sites (25 patients each site) with one CV risk factor will be randomised to either Q-risk 3 score or to screening CTCA.

DETAILED DESCRIPTION:
This is a pilot study- 50 patients, randomised 1:1 to each arm (25 patients per arm). This is 10% of the original sample size of 500. As this is a 2 centre study, each centre will recruit 25 patients and the financial requirement will be the responsibility of the individual centre.

Potential participants will be recruited from specialist non-Cardiology clinics in Sandwell and West Birmingham Hospitals (SWBH) NHS Trust and the Barts London hospital. Participants will be approached by members of the clinical care team when they attend the specialist non-Cardiology clinic. This study will be discussed with the participants and the patient information sheet handed over to them. Assent will be taken for further review in clinic by a member of the research team. Following this and written informed consent, they will be randomised to either CTCA or Q-risk 3 score.

Non-English-speaking patients will have a Trust translator (either language line or in-person).

Randomisation: Block randomisation with sealed envelope technique after written informed consent. Randomisation will be performed by members of the research team. Patients will randomised 1:1 to the interventional arm (CTCA) or Q-risk 3 score.

Blood tests: After consent, a routine blood sample of 20 millilitres (ml) - will be collected. The blood sample will be analysed at sites local lab and the following results will be collected: full blood count, urea and electrolytes, glycosylated haemoglobin (HbA1c), lipid profile and lipoprotein a (Lp (a) ).

Follow up: At one year from recruitment, patients will have a telephonic follow up to obtain information regarding occurrence of any events and/or hospitalisation.

Data collection, management and analysis:

* Electronic case record file (eCRF) and online database to collect demographic, medical history, CTCA report and Q risk score information.
* Blood samples in both groups
* Comparison of demographics, bloods, proportion started on primary prevention treatment between the CTCA and Q-risk 3 group.
* Categorical variables will be presented as percentage and compared with the chi square or Fisher's test.
* Continuous variables will be presented as mean (+/- standard deviation) and tested for normalcy by
* Kolmogorov-Smirnov test. Normal variables will be compared by student's t-test or in the case or non-normal variables by Analysis of Variance (ANOVA).
* Proportion of patients in the CTCA arm who receive primary prevention treatment versus proportion in the Q-risk arm who receive primary prevention treatment will be compared, as will the composite of event rates and hospital admissions at one year.
* In addition, the association of Q-risk 3 score with plaque on CTCA will be analysed by ROC curve.

Confidentiality: No identifiable data will be leaving the Trust. The respective sites (SWBH and Barts hospitals) will individually perform the CTCA and Q-risk 3 score on their cohort of patients and report it individually Authorised members of the Sponsor organisation will monitor the research at appropriate timelines and therefore have access to patients' identifiable information. Patients recruited will be allocated a participant ID.

Pseudonymised data will be collected on electronic case report forms (CRFs). Following completion of the study, anonymised data will be analysed. NHS indemnity will apply to this study. Study data will be stored for a maximum of 5 years after closure.

Ethics: All required ethical approval(s) for the trial will be sought using the Integrated Research Application System. The trial will be conducted in accordance with all relevant regulations.

Before enrolling patients into the trial, each trial site must ensure that the local conduct of the trial has the agreement of the relevant NHS Trust Research & Development (R&D) department. Sites will not be permitted to enrol patients into the trial until written confirmation of Capacity and Capability (CC&C) is received. All patients will be consented prior to inclusion in this study.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic South Asian patients of age

  * men≥30 years ≤60 years
  * Women >50 years ≤60 years

Plus at least one of the following risk factors:

* hypertension (HTN)
* diabetes mellitus (DM)
* hyperlipidaemia
* family history of premature coronary artery disease (male <45 years, female <55 years)
* smoking (current or ex-smoker in the last 3 months)

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded

  * Patients unable to give written informed consent
  * History of previous coronary events/CABG/ coronary stenting or CTCA in the last 4 years
  * Patients with pre-existing cardiac symptoms
  * Patients who could or are pregnant
  * Allergy to iodine contrast
  * Active ongoing malignancy and treatment for the same
  * eGFR ≤30ml/min/1.72m2
  * Participation in any other interventional research trial

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Patients treated by primary prevention | through study completion, an average of 1 year
  To compare the proportion of patients treated by primary prevention therapy with screening CTCA versus Q-risk 3 score

SECONDARY OUTCOMES:
Association of Q risk 3 score with plaque seen on CTCA | through study completion, an average of 1 year
  To assess the association of Q-risk 3 score with plaque on CTCA by receiver operating curve
Predictors of plaque on CTCA | through study completion, an average of 1 year
  To assess the predictors of plaque on CTCA by Cox proportional hazard analysis

CONTACTS AND LOCATIONS:
Overall Officials: Vinoda Sharma, FRCP FESC, Study Chair — Sandwell & West Birmingham Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No
This is a pilot study which will help to conduct larger studies which will confirm or refute the pilot study findings

REFERENCES:
- [Background] Lim MC, Wong TW, Yaneza LO, De Larrazabal C, Lau JK, Boey HK. Non-invasive detection of significant coronary artery disease with multi-section computed tomography angiography in patients with suspected coronary artery disease. Clin Radiol. 2006 Feb;61(2):174-80. doi: 10.1016/j.crad.2005.09.006. PMID 16439223
- [Background] Hughes DM, Coronado JIC, Schofield P, Yiu ZZN, Zhao SS. The predictive accuracy of cardiovascular disease risk prediction tools in inflammatory arthritis and psoriasis: an observational validation study using the Clinical Practice Research Datalink. Rheumatology (Oxford). 2024 Dec 1;63(12):3432-3441. doi: 10.1093/rheumatology/kead610. PMID 37966910
- [Background] Hippisley-Cox J, Coupland C, Brindle P. Development and validation of QRISK3 risk prediction algorithms to estimate future risk of cardiovascular disease: prospective cohort study. BMJ. 2017 May 23;357:j2099. doi: 10.1136/bmj.j2099. PMID 28536104
- [Background] Harding S. Mortality of migrants from the Indian subcontinent to England and Wales: effect of duration of residence. Epidemiology. 2003 May;14(3):287-92. PMID 12859028